CLINICAL TRIAL: NCT05578196
Title: Fecal Microbial Transplantation in Critically Ill Patients With Severe Infections:A Randomized Clinical Trial
Brief Title: Fecal Microbial Transplantation in Critically Ill Patients With Severe Infections.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Chen Yuanzhuo, associate chief physician, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMT20220925
Record Dates: First submitted 2022-09-25; First posted 2022-10-13 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Sepsis; Infections
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group with FMT (Experimental): The gastrointestinal tube access was established, and the standard preparation of fecal bacteria solution 20ml (frozen at -80 ° C, melted at room temperature before use) was injected through the gastrointestinal tube once a day for 6 consecutive days. The other treatment measures were the same as those of the control group
  Interventions: Drug: fecal bacteria solution
- The control group with physiological saline (Other): The gastrointestinal tube access was established, and the standard preparation of physiological saline solution 20ml
  Interventions: Drug: physiological saline solution

INTERVENTIONS:
Drug: fecal bacteria solution — The gastrointestinal tube access was established, and the standard preparation of fecal bacteria solution 20ml (frozen at -80 ° C, melted at room temperature before use) was injected through the gastrointestinal tube once a day for 6 consecutive days. The other treatment measures were the same as those of the control group.
  Arms: The experimental group with FMT
Drug: physiological saline solution — physiological saline solution 20ml
  Arms: The control group with physiological saline

SUMMARY:
Fecal microbial transplantation is to transplant functional microbiota from the feces of healthy people into the gastrointestinal tract of patients, reconstruct new intestinal microbiota, and realize the treatment of intestinal and extra-intestinal diseases. Compared with ordinary commercial probiotics, FMT is more consistent with the composition of the intestinal microecological structure and can recover intestinal flora to the maximum extent and faster. FMT increases intestinal bacteria production function and helps to restore the systemic immune response so that sepsis pathogens are removed. The aim of this trial was to investigate the clinical effect of FMT in the treatment of patients with severe infections.

DETAILED DESCRIPTION:
The gastrointestinal tube access was established, and the standard preparation of fecal bacteria solution 20ml (frozen at -80 ° C, melted at room temperature before use) was injected through the gastrointestinal tube once a day for 6 consecutive days. The other treatment measures were the same as those of the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe infections, which is infected patients SAFA≥2 OR APACHE Ⅱ≥15
* Aged ≥14 years
* Patients or their family members agreed to participate in this study

Exclusion Criteria:

* Advanced tumors or diseases associated with systemic immunosuppression
* Pregnant women
* Patients with severe intestinal ulcer or perforation
* Unable to complete oral administration and no effective artificial feeding pipeline.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-09-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | up to 28 days in ICU
  Clinical outcome

SECONDARY OUTCOMES:
Gut microbiota distribution assessed by 16SrDNA | up to 6 days after fecal microbial transplantation
  16SrDNA

CONTACTS AND LOCATIONS:
Overall Officials: YuanZhuo Chen, Study Chair — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haak BW, Prescott HC, Wiersinga WJ. Therapeutic Potential of the Gut Microbiota in the Prevention and Treatment of Sepsis. Front Immunol. 2018 Sep 10;9:2042. doi: 10.3389/fimmu.2018.02042. eCollection 2018. PMID 30250472